CLINICAL TRIAL: NCT07315230
Title: Pediatric Midline Post Fossa Tumors Prognostic Factors and Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Abdelaziz Hassan, Resident at Neurosurgery Department, Assiut University, Assiut University
Other Study IDs: Midline posterior fossa tumors
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Tumor; Midline Posterior Fossa Tumors
Keywords: Pediatric; Midline Posterior Fossa Tumors; Prognostic factors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will follow children younger than 18 years with midline posterior fossa brain tumors who undergo standard surgical resection at Assiut University Hospital. The aim is to evaluate functional outcome using the modified Rankin Scale and to explore how tumor type, extent of resection, and perioperative factors are associated with postoperative morbidity and survival. Results may help improve risk stratification and guide individualized treatment strategies for pediatric patients with these tumors.

DETAILED DESCRIPTION:
This is a single-center, prospective, hospital-based observational cohort study conducted in the Neurosurgery Department at Assiut University Hospital. Consecutive pediatric patients (<18 years) with radiologically confirmed midline posterior fossa tumors who are considered fit for surgery will be enrolled after informed consent from parents or legal guardians. Preoperative assessment will include demographic data, clinical presentation, neurological examination, and standardized brain MRI.

All patients will undergo surgical resection according to routine neurosurgical practice, using an operating microscope and standard approaches appropriate to tumor location. Intraoperative details (position, approach, estimated blood loss, complications, and surgeon-assessed extent of resection) will be recorded, and tumor specimens will be sent for histopathological diagnosis. Early postoperative evaluation will document Glasgow Coma Scale, intensive care and hospital stay, and complications such as cerebellar mutism, hydrocephalus, and cranial nerve deficits.

Postoperative imaging (CT or MRI) within 48 hours will be used to classify the extent of resection as gross total, near total, subtotal, or partial. Functional outcome will be assessed using the modified Rankin Scale at approximately 6 months after surgery, with patients categorized as having good (mRS 1-3) or poor (mRS 4-6) outcome. Additional follow-up visits (for example at 3 months, 6 months, and annually when feasible) will document tumor recurrence, need for adjuvant therapies, and long-term neurological sequelae.

The main objective is to evaluate functional and radiological outcomes after surgical management of pediatric midline posterior fossa tumors and to identify prognostic factors that influence morbidity, mortality, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients less than 18 years old
* patient with midline posterior fossa tumors
* patient is fit for surgery

Exclusion Criteria:

* patinent older than 18 years old
* patients with non-midline posterior fossa or other brain tumors.
* patient is unfit for surgery .
* Incomplete Data: Missing essential study data.
* Secondary Malignancy: Metastatic disease.

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients younger than 18 years presenting to the Neurosurgery Department, Assiut University Hospital, with radiologically confirmed midline posterior fossa brain tumors and considered candidates for surgical resection. Participants are recruited consecutively from routine clinical care and followed postoperatively for functional and radiological outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome After Surgical Resection of Pediatric Midline Posterior Fossa Tumors | 6 months after surgery.
  Assessment of the patient's functional status using the modified Rankin Scale (mRS) after surgical resection of a midline posterior fossa tumor in children, categorized as good outcome (mRS 1-3) or poor outcome (mRS 4-6).